CLINICAL TRIAL: NCT02715219
Title: The Effect of an Asthma Education Programme on Patient's Knowledge Regarding Asthma Disease and Inhaler Technique: Randomized Control Trial
Brief Title: The Effect of an AEP on Patient's Knowledge Regarding Asthma Disease and Inhaler Technique: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Lilyiana Binti Pengui, Principal investigator, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMRR-14-1642-23836
Record Dates: First submitted 2016-02-25; First posted 2016-03-22 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): Subjects in intervention group will be given an appointment date to attend the an Asthma Education Programme.
  Interventions: Other: Asthma Education Programme
- control group (No Intervention): Subjects in control group will routinely go for the normal follow up in Respiratory Clinic without receive any intervention.

INTERVENTIONS:
Other: Asthma Education Programme — The Asthma Education Programme consists of four items. 1. Education video for Asthmatic patient adapted from Info Sehat by Bahagian Pendidikan Kesihatan Kementerian Kesihatan Malaysia which is explaining about Asthma disease, medication and patient responsibility in Asthma management. 2. Small group discussion with subject's to help them understand better in Asthma management. 3. Face to face demonstration and teaching of inhaler technique by three trained nurse in small group range of two to five subjects. At the end of the AEP subject will received a 4. Pamphlet will be obtain from Patients' Education Unit in Ampang Hospital containing vital information about Asthma disease and management. The intervention estimated will take 1 hour to 1 hour 30 minutes to be completed.
  Arms: intervention group

SUMMARY:
Asthma is an important chronic disease that causes a significant public health problem and the commonest medical conditions treated in health clinics giving rise to considerable morbidity and mortality. Several studies suggested that improvement of patient knowledge has become a key component of asthma management. In the study setting the education material for Asthma patient is available however the proper cannel to deliver it to patient remains a puzzle to the researcher, therefore this study is trying to close the gap between Asthma education material and patient.The aim of the study is to investigate the effectiveness of an Asthma Education Program (AEP) result in improvement of patient's knowledge, medication adherence and inhaler technique.This is an experimental study a clinical trials. Data will be gathered utilising three an adapted instrument to assess patient knowledge of their disease, medication adherence and inhaler technique. Patients who are came to Asthma Bay in Emergency Department, Respiratory Clinic for routine follow up and admitted to ward will be recruited as study subjects. Subject who are agree to enrol in the study will be randomized into intervention and control group. Subjects in intervention group will be undergone one session of an AEP, however there are no intervention for control group but continue routinely follow up in Respiratory Clinic. To obtain the study result descriptive and inferential statistical analysis will be performed. To analyse the statistical significant of the change in patients' health outcome the pre and post of AEP independent t-test or chi-square test will be used.The expected finding of this study is to determine the effectiveness of AEP result in of patients' knowledge regarding asthma disease, medication adherence and inhaler technique, pre and post of AEP.

Keywords: asthma, asthma education program.

DETAILED DESCRIPTION:
Asthma is an important chronic disease and a significant public health problem. Prevalence of asthma is on the rise in all regions of the world, affecting all ages but more commonly among children.The burden and suffering caused by chronic respiratory disease has been identified by the World Health Organization (WHO) as a priority. In Malaysia, asthma is among the commonest medical conditions treated in health clinics giving rise to considerable morbidity and mortality (Bahari, Mohd Nur & Rahman, 2003).Much of the morbidity from asthma is believed to be due to factors such as denial of having a chronic condition (GINA, 2002), poor knowledge of the disease process and medication use (Gibson et al., 2004) , poor understanding on the use of inhalers (Thapar, 1994) and poor self-management (Wilson et al., 1993; Hilton, Sibbald, Anderson & Freeling, 1986). Patient education is becoming an essential area of service provision, with our increasing population of people with chronic diseases and conditions requiring long-term management in the community. Inadequate patient education has been cited as a potential cause of re-attendance and the optimal format of education is uncertain. Numerous studies worldwide have evaluated the impact of patient education and indicated that each of the above components is amenable to asthma education (GINA, 2002). Thus, patient education has become a key component of asthma management for asthma patients at all age groups (Lai, et al., 2002; Harrison, 1998). Despite the means to control asthma effectively, many asthma sufferers in Malaysia are not availing themselves of such strategies, leading to avoidable problems that can range from frequent asthma attacks to even death in certain circumstances. Much of the morbidity from asthma is believed to be due to factors such as denial of having a chronic condition (Gibson, et al., 2004), poor knowledge of the disease process and medication use (Thapar, 1994), poor understanding on the use of inhalers (Wilson, et al., 1993) and poor self-management (Lai, et al., 2002; Hilton, Sibbald, Anderson & Freeling, 1986). However the effectiveness of patient education for asthma in a hospital-based setting in Malaysia has not been previously evaluated and remains a puzzle to the researcher. With the concern the researcher would like to explore the effectiveness of Asthma Education Programme in improvement of patients' knowledge regarding asthma, medication adherence and inhaler technique.

Research question. Does an Asthma Education Programme result in improvement of patient's knowledge regarding asthma disease and inhaler technique?

Research aims. i. To compare patient knowledge regarding asthma disease between intervention and control group . ii. To compare patient inhaler technique between intervention and control group. iii. To assess the association between patient's demographic data and health outcomes (Knowledge and inhaler technique).

Study design. This is an experimental study a clinical trials. The period of this study is six month which is start from July 2015 to January 2016.

Study Setting This study will be conducted in Ampang Hospital a government public tertiary specialist hospital in Ampang, Selangor Malaysia.

Population (N). Asthmatic patients who treated in Ampang Hospital during the study period.

Target Population. Asthmatic patients who will be presented in Asthma Bay, Respiratory Clinic or who are admitted to general medical wards for uncontrolled acute asthma attack.

Sample Size (n). The sample size of the study calculated using formula of hypothesis testing for difference in proportions and the researcher determine effect size of 15% as significant change, so the study need at least 129 subjects in each of arm.

Inclusion Criteria.

* Patient above age of 18 years.
* Have confirmed diagnosis of bronchial asthma in the medical record.
* Have used inhaler medication past 1 year.

Exclusion Criteria.

- Patient with significant medical comorbidity such as heart disease, chronic obstructive pulmonary disease, chronic renal disease, stroke, psychiatric problem or inability to follow instruction.

Sampling method. Patients who are presented in Asthma Bay, Respiratory Clinic and been admitted to general medical ward and fulfil the inclusion criteria will be recruited to be subject of the study. Patients' will be given an explanation about the study and written consent will be obtained who are agreeing to participate in the study. Patients will be randomized using simple computer randomization.

Instrument. The data for the study will be collected utilizing three adapted instrument from previous study and the permission to use the questionnaire will be obtained through email.

Questionnaire (Part A) : Demographic data Part A consist of information about subjects demographic data, such as age, sex, race, education level, history of childhood asthma and number of ward admission or ED visits in the past one year. In the post test questionnaire this part will be omitted but the subsequent layouts were similar.

Questionnaire (Part B) : Asthmatic patients' knowledge about their disease. Part B consists of twenty close ended question, to assess respondents' basic knowledge on their disease, medication and treatment maintenance. The questionnaire adapted from previous study by Baez Saldana, et.al (2007). Responses will be made on selection of three choice of answer which is "a", "b" or "c".

Questionnaire (Part C) : Multiple checklist of inhaler technique. To evaluate the respondents' inhaler technique a single page with multiple checklist created by Vicky Kritikos will be adapted. The checklists contain six types of inhaler technique medication, such as Metered Dose Inhaler (MDI) with spacer, MDI, Turbuhaler, Accuhaler, Intranasal device and Handihaler. Subjects will be asked by investigator to demonstrate how they use the inhaler medication individually. Incorrect step of inhaler technique will be highlighted and emphasis during the AEP.

Validity and Reliability. The validity and reliability of instruments content will be checked by expertise panel such as a respiratory physician and pilot study will be held for test-retest and Cronbach alpha test.

Data Collection. There are three phases involve in data collection of this study. Following Ethic Committee approval the researcher will meet up with Head Department of Emergency Department, Medical and respiratory physician in charge of Respiratory Clinic to notify them about the study and formal letter explaining the purpose of the study and copy of ethical approval will be given to them.

Phase 1: Recruitment and randomization. Patients who are fullfill the subjects inclusion criteria in those units will be approached and subject will be given briefly explanation about the study and written consent will be obtained. Subjects (single blind study) will be randomized using simple computer randomization. Subjects in intervention group will be given an appointment date to attend the an Asthma Education Programme and subjects in control group will routinely go for the normal follow up.

Phase 2: Baseline data collection and AED session for intervention group. Baseline data collection for subject in control group will be held in wards or Respiratory Clinic and for subject recruited from Asthma Bay the baseline data will be collected during their routine follow up in Respiratory Clinic. Upon completion collection of baseline data subject will be given appointment date 4 weeks or same day clinic visit for second session of data collection. For intervention group the baseline data collection will be held prior to Asthma Education Programme and appointment date will be given after 4 weeks for second data collection.The Asthma Education Programme consists of four items.

1. Education video for Asthmatic patient adapted from Info Sehat by Bahagian Pendidikan Kesihatan Kementerian Kesihatan Malaysia which is explaining about Asthma disease, medication and patient responsibility in Asthma management.
2. Small group discussion with subject's to help them understand better in Asthma management.
3. Face to face demonstration and teaching of inhaler technique.
4. Pamphlet will be given to subjects which is prepared by Bahagian Pendidikan Kesihatan Kementerian Malaysia containing vital information about Asthma disease and management.

Phase 3: Second data collection, After four weeks collection of the baseline data, both group of subjects who are attending follow-up in Respiratory Clinic or by appointment given by the researcher will be required to answer the same questionnaire and demonstrate their inhaler technique.

Data Analysis The collected data will be reviewed by researcher and cross-check by two independent individuals. The data will be entered into Statistical Package for Social Science (SPSS) version 20 and will be analysed using descriptive and inferential statistical. Questionnaire Part A will be analysed using frequency and mean statistical, the result will be displayed in tables.To analyse the association between subjects' demographic data and knowledge status and inhaler technique Chi-square test or independent t-test will be used. Part B of the questionnaire containing of 20 items asking regarding respondents' knowledge of their disease, medication and treatment maintenance. ". Responses will be made on a three choice of answer. Each of the correct answer will be given scores 1, and 0 scores for wrong answers. Researchers will determined the status of respondents' knowledge in two categories, which is the total score from 15 to 20, is in category of good knowledge and total score from one to 14 is in poor knowledge category. In order to obtain result descriptive statistic (mean(SD) analysis will be performed. For result comparison between statistic (mean (SD) analysis will be performed. For result comparison between intervention and control group Independent t- test analysis will be used. Part C of the questionnaire is to evaluate the respondents' inhaler technique using a single page with multiple types of inhaler technique checklist such as Metered Dose Inhaler (MDI), MDI with spacer, Turbuhaler, Accuhaler, Intranasal device and Handihaler.

Ethical Considerations The study is registered and approved by National Medical Research Register, Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of bronchial asthma in the medical record.
* Have used inhaler medication past 1 year.

Exclusion Criteria:

* Patient with significant medical comorbidity
* heart disease
* chronic obstructive pulmonary disease
* chronic renal disease
* stroke
* psychiatric problem or inability to follow instruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The difference of subjects' knowledge score as assessed using a questionnaire. | 4 weeks
  To compare patient knowledge status regarding asthma disease between two groups .

SECONDARY OUTCOMES:
The difference of patient inhaler technique status as assessed using a checklist. | 4 weeks
  To compare patient inhaler technique between two groups.
The association between patient's demographic data and knowledge status, medication adherence and inhaler technique. | 4 weeks.
  To compare the association result between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lilyiana Pengui, nursing, Principal Investigator — Clinical Research Centre, Malaysia

IPD SHARING:
Plan to Share IPD: Yes